CLINICAL TRIAL: NCT06845631
Title: Retrospective-Prospective Clinical Trial Investigating the Treatment of Chronic Pain With the Freedom Peripheral Nerve Stimulation System
Brief Title: Retrospective-Prospective PNS Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Curonix LLC (Industry)
Collaborators: MetroHealth System, Ohio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P011
Record Dates: First submitted 2025-02-11; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: chronic pain, PNS, Retrospective, prospective
MeSH Terms: conditions — Chronic Pain | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Retrospective/Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Observational (Experimental): observational
  Interventions: Device: PNS device, observational study, no intervention during study

INTERVENTIONS:
Device: PNS device, observational study, no intervention during study — PNS device, observational study, no intervention during study

SUMMARY:
This is a retrospective-prospective study in which 40 patients have received a permanent Freedom PNS System. Subjects presented with chronic, intractable pain of peripheral nerve origin refractory to standard medical and/or surgical treatment.

A retrospective chart review will be conducted to assess baseline and follow-up parameters in patients who have received a permanent implant with the Freedom PNS system for at least 12 months. Missing data might be collected after informed consent.

ELIGIBILITY:
Inclusion Criteria:

A. Subject is ≥ 18 years of age at time permanent implant; B. Subject has been implanted with the Freedom PNS system; C. Subject is willing to attend visit as scheduled, and comply with the study requirements (if prospective); D. Patient is capable of giving informed consent.

Exclusion Criteria:

A. Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study while participating in this study (if prospective); B. Any additional active implanted devices for the treatment of chronic pain in addition to the Freedom PNS system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 12 months
  A text description of the subject's pain location(s) and severity will be recorded to correlate with subject feedback. The VRS will be used to measure severity.

SECONDARY OUTCOMES:
Opioids | 12 months
  Each subject's opioid medication type, dose, frequency, and method of administration will be recorded at baseline and follow-up visit.
Work status | 12 months
  Work history and status will be evaluated based on a subject's self-reported questionnaire(s) completed at screening/baseline and all follow up visits.
GPES | 12 months
  Subject satisfaction with the implant will be measured by assessing global perceived effects (GPES) on a 7-point scale (1 = worst and 7 = best)
Amount of sleep | 12 months
  Average hours of sleep per night will be evaluated at baseline and all follow-up visits
Sleep disturbances | 12 months
  The amount of sleep disturbances (awakenings) per night to track quality of sleep
EQ-5D-5L | 12 months
  The European Quality of Life - 5 Dimension - 5L (EQ-5D-5L) is a standardized instrument for use as a measure of health outcome.
Claims data | 12 months
  The value of claims data at the site will be measured from 1 year before and up to the date of implant and compared to the claims value up to 1 year after implant. The number of appointments will be collected together with the CPT codes used for pain interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Metrohealth System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided